CLINICAL TRIAL: NCT06457880
Title: Pericapsular Nerve Group (PENG) Block vs Femoral Nerve Block (FNB) + Obturator Nerve Block (ONB) in Patients Undergoing Hip Fracture Surgery With Contraindications to Neuraxial Anesthesia
Brief Title: PENG Block vs FNB + ONB in Patients Undergoing Hip Fracture Surgery With Contraindications to Neuraxial Anesthesia
Acronym: PENG/FNB+ONB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Francesca Gargano, Medical director, Anesthesiologist, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Campus Bio-Medico
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hip Fractures; Pain, Postoperative; Coagulopathy; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative; Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block (Experimental): Before surgery, Patients undergo to ultrasound guided PENG block administering ropivacaine 0.5 % 20 mL.
  Interventions: Procedure: PENG BLOCK
- Femoral nerve block + Obturator nerve block (Active Comparator): Before surgery, Patients undergo to ultrasound guided femoral nerve block (ropivacaine 0.5 % 15 mL) + obturator nerve block (ropivacaine 0.5% 5 mL).
  Interventions: Procedure: Femoral Nerve Block; Procedure: Obturator Nerve Block

INTERVENTIONS:
Procedure: PENG BLOCK — Preoperative ultrasound guided PENG block (ropivacaine 0.5 % 20 mL)
  Arms: PENG block
Procedure: Femoral Nerve Block — Preoperative ultrasound guided femoral nerve block (ropivacaine 0.5 % 15 mL)
  Arms: Femoral nerve block + Obturator nerve block
Procedure: Obturator Nerve Block — Preoperative ultrasound guided obturator nerve block (ropivacaine 0.5 % 5 mL)
  Arms: Femoral nerve block + Obturator nerve block

SUMMARY:
The aim of the study is to demonstrate the efficacy of PENG block as the main anesthetic technique to manage perioperative analgesia for hip fracture surgery compared to femoral and obturator nerve block in patients with contraindications to spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo hip surgery
* patients with contraindications at spinal anesthesia

Exclusion Criteria:

* allergy at local anesthetic
* age under 18 or weight under 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
preoperative pain | 30 minutes
  Preoperative pain score expressed by numerical rating scale 0-10
Pain following regional anesthesia | 30 minutes
  Preoperative pain score following regional anesthesia execution expressed by numerical rating scale 0-10
Postoperative pain | 24 hours
  Postoperative pain score expressed by a numerical rating scale 0-10

SECONDARY OUTCOMES:
Morphine milligrams (mg) consumption | 24 hours
  needed opioid rescue therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Bio Medico, Roma, Italy